CLINICAL TRIAL: NCT01437150
Title: Treatment of Acetabular Posterior Wall Fracture With Anatomical Locking Plate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peifu Tang (Other)
Responsible Party: Sponsor-Investigator, Peifu Tang, Chief, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLAGH OD 11
Record Dates: First submitted 2011-09-01; First posted 2011-09-20 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Fracture of Acetabulum
Keywords: surgery; fixation; bone plate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simple posterior wall fracture (Experimental): Simple posterior wall fracture means the fracture was only occurred in the posterior wall of acetabular.
  Interventions: Device: Anatomical locking plate; Procedure: The Reconstructive Plate
- Complex posterior wall fracture (Experimental): Complex posterior wall fracture means the fracture was not only occurred in the posterior wall of acetabular, but also occurred in other part of acetabular.
  Interventions: Device: Anatomical locking plate; Procedure: The Reconstructive Plate

INTERVENTIONS:
Device: Anatomical locking plate — This is a new fixation treat for acetabular posterior wall fracture.
  Other Names: WEIGAO ORTHOPAEDIC DEVICE CO.LTD.; ZL200920105202.7
Procedure: The Reconstructive Plate — Reconstructive plate was used very common in treatment of acetabular fracture.
  Other Names: The Reconstructive Plate System

SUMMARY:
The purpose of this study is to determine whether this new anatomical locking plate is more effective and easy to operate than other plate in the treatment of acetabular posterior wall fracture.

DETAILED DESCRIPTION:
Acetabular fractures were very common in high-energy injury, because of the anatomic of acetabular was in deep location and the complex form cause the diagnosis and treatment was difficult. For most of displaced acetabular fractures, the preferred treatment is open reduction and internal fixation. The purpose of surgery is to restore acetabular integrity and stability, allow early exercise, decrease complication. Acetabular posterior wall fractures were the most common, the current clinical application fixation of acetabular fractures were common plate and reconstruction steel plate. But when the acetabular posterior wall was fracture, some patients were not satisfied after surgery. The reason is mainly because the reconstruction plate need remoulding in surgery, and it not only led to the extension of operation time, but also cause poor attach. Otherwise, the reconstruction plate need location the angle of screw in surgery. If the operator lack of experience will make into the harm surrounding vessels and nerves. Some research has achieved the improvement from the anatomy of acetabular fractures in the locking plate. But there is not any plate match with the anatomy of the acetabular posterior wall.

This anatomical bone plate was designed base on before plate and had patent protection which is used in clinical trial. It was a new type of internal fixation of acetabular posterior wall fracture, this plate improve the shortcomings of existing technology, provides a pre-formed anatomical fixation plate , the direction of the locking screw holes. This design provide a better attach of acetabular posterior wall, more safe use the screw, making more stable and reliable fixation. This fixation plate was not only suitable for an experienced doctor, but also suitable for a less experienced doctors in theory. They can quickly and accurately fixed in its correct position, thus this fixation plate have advantages of improve surgical success rates, shorter hospital stay, reduce disease painful and it can used in all adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18 years and older (with no upper age limit).
* Fracture of the acetabular posterior wall fracture confirmed with either anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
* Operative treatment of fractures within 14 days of presenting to the emergency room.
* Patient was ambulatory prior to fracture, though they may have used an aid such as a cane or a walker.
* Anticipated medical optimalization for operation.
* Provision of informed consent by patient or legal guardian.
* No other major trauma.

Exclusion Criteria:

* Refuse to participate.
* Patients not suitable for internal fixation (i.e., severe osteoarthritis, rheumatoid arthritis, or pathologic fracture).
* Associated major injuries of the lower extremity (i.e., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula, knee, or femur; dislocations of the ankle, knee, or hip; or femoral head defects or fracture).
* Retained hardware around the affected acetabular.
* Infection around the acetabular (i.e., soft tissue or bone).
* Patients with disorders of bone metabolism except osteoporosis (i.e., Paget's disease, renal osteodystrophy, osteomalacia).
* Moderate or severe cognitively impaired patients (i.e., Six Item Screener with 3 or more errors).
* Patients with Parkinson's disease (or dementia) severe enough to increase the likelihood of falling or severe enough to compromise rehabilitation.
* Likely problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Bone healing condition | six months
  Bone healing condition was checked by radiological examination.

SECONDARY OUTCOMES:
Rates of revision surgery | one year
Patient quality of life | one year
  SF-36, ADL, FIM
Complications | one year
  mortality, nonunion, implant breakage/failure, infection, DVT

CONTACTS AND LOCATIONS:
Overall Officials: Tang Peifu, Dr., Study Chair — Chinese PLA General Hospital
Locations (1):
- Orthopedics department; The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality, China